CLINICAL TRIAL: NCT02026297
Title: The Influence of Prophylactic Tranexamic Acid on Thromboelastography During Cesarean Delivery: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Tranexamic Acid and Thromboelastography During Cesarean Delivery
Acronym: TA TEG
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding and manpower unavailable, completion within a reasonable timeframe not possible.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Michaela Kristina Farber, MD, Instructor of Anesthesia, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2013P002452
Record Dates: First submitted 2013-12-22; First posted 2014-01-01 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Postpartum Hemorrhage
Keywords: postpartum hemorrhage; estimated blood loss; coagulation; thromboelastography; tranexamic acid
MeSH Terms: conditions — Postpartum Hemorrhage; Thrombosis | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control, low risk PPH (Placebo Comparator): Patients at lower risk for postpartum hemorrhage during cesarean delivery, to receive standard of care NOT including tranexamic acid.
  Interventions: Drug: Placebo; Normal Saline
- Treated, low risk PPH (Experimental): Patients at lower risk for postpartum hemorrhage during cesarean delivery, to receive standard of care AND tranexamic acid.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — 1 gram IV over 10 minutes
  Arms: Treated, low risk PPH
Drug: Placebo; Normal Saline — 0.9% Normal Saline
  Arms: Control, low risk PPH

SUMMARY:
The aim of this study is to characterize the coagulation changes, using thromboelastography (TEG), after prophylactic tranexamic administration during cesarean delivery. Specifically, TEG values will be compared in patients who receive prophylactic tranexamic acid or placebo before surgery, during elective cesarean delivery, and 2 hours postpartum.

Postpartum hemorrhage (PPH) is increasing in incidence in the United States, renewing interest in multimodal approaches to blood conservation during cesarean delivery. Pharmacologic therapy with the antifibrinolytic agent, tranexamic acid (TA), has been shown to reduce estimated blood loss (EBL) during cesarean delivery, but its effect on global coagulation as assessed by TEG, and how this correlates with lowering blood loss, has not been elucidated.

This study will be conducted as a randomized, double-blind, controlled trial with two study arms: control (60 patients); and treatment (60 patients).

Subjects will be pre-medicated with routine pre-cesarean delivery medications including oral sodium citrate 30 mL and intravenous (IV) metoclopramide 10 mg. A peripheral IV and noninvasive hemoglobin monitor will be placed, and baseline labs sent: type and screen, serum hemoglobin, platelet count, fibrinogen, activated partial thromboplastin time (aPTT), prothrombin time (PT), and baseline TEG values (r time, k time, alpha angle, and maximum amplitude). Patients will have blood pressure, heart rate, and pulse oximetry measured throughout surgery as per standard of care. Patients will all receive IV lactated Ringers' (LR) solution prior to surgery and throughout surgery, with volume recorded and a goal of less than 2 L unless more IV fluid is clinically indicated. All patients will have a spinal anesthetic as per standard of care, with hyperbaric bupivacaine 12 mg, fentanyl 10 μg, and hydromorphone 100 μg. If the anesthetic plan is altered (combined spinal-epidural, general anesthesia conversion, general anesthesia planned), indications and medication doses used will be noted for analysis.

Immediately following induction of anesthesia and prior to skin incision, infusion of study solution will be initiated.

Study solutions will consist of:

1. Control group: 100 mL 0.9% normal saline (NS).
2. Treatment group: 100 mL 0.9% NS containing 1g tranexamic acid (TA). Study solution will be infused via an infusion pump over 10 minutes. Blood loss will be measured by visual estimate and weight of surgical sponges. Noninvasive hemoglobin will be measured throughout the study. All routine care lab values will be noted. At minimum, one lab panel will be sent one hour after study solution initiation (hemoglobin, fibrinogen, platelet count, aPTT, PT, and TEG).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class I or II
* aged 18-50 years
* singleton vertex pregnancy
* scheduled elective cesarean delivery (with or without prior labor) with a planned pfannenstiel incision

Exclusion Criteria:

* allergy to tranexamic acid
* history of inherited or acquired thrombophilia
* history of deep vein thrombosis or pulmonary embolism, or use of anticoagulant medication.
* preeclampsia, hemolysis, elevated liver enzymes, low platelet syndrome
* seizure disorder

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2020-02-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control, Low Risk PPH | Treated, Low Risk PPH
Started | 7 | 13
Completed | 7 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients scheduled for elective cesarean delivery with low risk for postpartum hemorrhage.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control, Low Risk PPH | Treated, Low Risk PPH | Total
Number analyzed (Participants) | 7 | 13 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 13 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 35.2 [30 to 40] | 31.9 [20 to 39] | 32.9 [20 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 20
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 13 | 20

OUTCOME MEASURES:

1. Primary Outcome: TEG Value- Thromboelastography R-time, Control and Treated Groups
Description: Blood samples will be collected for evaluation one our after initiation of the study infusion. Whole blood samples are tested in a point-of-care thromboelastography machine and R time, or time to initiation of clot formation, is measured in minutes.
Time Frame: one hour after initiation of study infusion
Population: Thromboelastography R-time
Measure: Mean (Inter-Quartile Range); unit: minutes
Arm/Group | Control, Low Risk PPH | Treated, Low Risk PPH
Number analyzed (Participants) | 7 | 13
minutes | 5.3 [4.2 to 7.7] | 4.2 [3.4 to 6.0]

2. Primary Outcome: Intraoperative Blood Loss
Description: Blood loss will be measured using the following methods:
  * visual estimate of blood in the suction canister
  * weight of surgical sponges
  * postoperative hemoglobin values
Time Frame: during surgery in the operating room
Population: weight of surgical sponges
Measure: Mean (Standard Error); unit: milliliters
Arm/Group | Control, Low Risk PPH | Treated, Low Risk PPH
Number analyzed (Participants) | 7 | 13
milliliters | 637 (151) | 685 (155)

3. Primary Outcome: Delayed Complications at the 6-Week Postpartum Visit With the Obstetrician.
Description: The electronic patient record from each patients' 6-week postpartum visit will be reviewed for the following:
  * delayed bleeding complications, defined as obstetric bleeding requiring surgical intervention, blood transfusion, or both.
  * thrombotic complications including: venous thrombus seen on ultrasound, thromboembolic event
Time Frame: 6 weeks postpartum
Population: postpartum Obstetrician evaluation at 6 weeks: obstetric bleeding requiring surgical intervention, blood transfusion, or both; thrombotic complications including: venous thrombus seen on ultrasound, thromboembolic event
Measure: Number; unit: complications
Arm/Group | Control, Low Risk PPH | Treated, Low Risk PPH
Number analyzed (Participants) | 7 | 13
complications | 0 | 0

ADVERSE EVENTS:
Time Frame: All patients enrolled in this study were evaluated in the immediate treatment period through the time of discharge (average duration 4 days) and then records were reviewed from the 6-week postpartum followup for delayed complications.
Description: * obstetric bleeding requiring surgical intervention, blood transfusion, or both.
  * thrombotic complications including: venous thrombus seen on ultrasound, thromboembolic event
Arm/Group | Control, Low Risk PPH | Treated, Low Risk PPH
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/13
Other Adverse Events (participants affected / at risk) | 0/7 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No